CLINICAL TRIAL: NCT02353403
Title: Postprandial Glycaemic and Insulinaemic Responses After Consumption of Dairy Desserts Containing Fructo-oligosaccharides in Adults.
Brief Title: Glycaemic and Insulinaemic Responses After Consumption of FOS.
Acronym: GLYCOFOS-cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Collaborators: Syral (Industry)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, MD, Endocrinologist, Nutritionist, Institut Pasteur de Lille
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2013-A00786-39
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Glycaemia
Keywords: Fructo-oligosaccharides; Sugar-reduced foods; Postprandial glucose response
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar (Placebo Comparator): Control group consuming a dairy dessert containing 35g of dextrose.
  Interventions: Other: Sugar
- FOS (Experimental): Group consuming a dairy dessert in which 30% of the dextrose was replaced by FOS.
  Interventions: Other: FOS

INTERVENTIONS:
Other: Sugar — A 210g chocolate dairy dessert made with 35g of dextrose.
  Arms: Sugar
Other: FOS — A 210g chocolate dairy dessert made with 24g of dextrose and 11.2g of FOS.
  Arms: FOS

SUMMARY:
The study aims to evaluate the glycaemic and insulinaemic response of short-chain fructo-oligosaccharides (scFOS) used to replace sugars (e.g. dextrose) in foods.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 25.0 kg/m² (included)
* Ready to keep the same volume of physical activity and the same dietary habits during the study and particularly 24 hours before each visit
* Be used to have breakfast
* Non-smoker for at least 3 months
* For the female participant: not being pregnant or breastfeeding and using efficient birth control
* Signed the consent form
* Able to follow the instructions of the study
* Health insured
* Accepted to be included in the National Registry for biomedical research Volunteers (Fichier VRB, Volontaires Recherches Biomédicales).

Exclusion Criteria:

* Fasting blood glucose over 6.1 mmol/L (1.10 g/L) (or diabetes treated or not)
* Fasting blood cholesterol over 6.35 mmol/L
* Fasting blood triglycerides over 1.70 mmol/L (or history of insulinoma)
* Fasting blood insulin under 20 mU/L
* Fasting HbA1c under 7%
* History of hypercholesterolemia, hypertension, diabetes or glucose intolerance treated or not
* History of dietary allergies or coeliac disease
* History of digestive system disease susceptible to modify digestion or absorption like Crohn's disease
* Somatic or psychiatric disorders
* Renal insufficiency (kidney failure)
* SGOT or ALAT over 52.5 U/L
* Smoker
* Consuming more than 3 alcoholic beverage a day
* Weight varied 3 kg the last 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Glycaemic response | 2 hours and 5 minutes
  Blood glucose kinetics with 7 points. Analysis of the Area under the curve of glucose.

SECONDARY OUTCOMES:
Insulinaemic response | 2 hours and 5 minutes
  Blood insulin kinetics with 7 points. Analysis of the Area under the curve of insulin.
Blood glucose peak (Cmax) | One-time data (the highest one) within the 2hrs 5mins kinetics.
  Peak of blood glucose during kinetics.
Blood insulin peak (Cmax) | One-time data (the highest one) within the 2hrs 5mins kinetics.
  Peak of blood insulin during kinetics.
Glucose Tmax : time to reach the peak of blood glucose | One time within the 2hrs 5mins kinetics.
Insulin Tmax : time to reach the peak of blood insulin | One time within the 2hrs 5mins kinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lecerf, MD, Principal Investigator — Institut Pasteur de Lille
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France